CLINICAL TRIAL: NCT04866680
Title: Personalized Circulating DNA Follow-up in Melanoma
Brief Title: Personalized Circulating DNA Follow-up in Melanoma (PERCIMEL)
Acronym: PERCIMEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01904-39
Record Dates: First submitted 2021-03-09; First posted 2021-04-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Melanoma
Keywords: Circulating tumour DNA; immunotherapy; targeted therapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Circulating DNA follow-up (Experimental): FFPE tissue sample + blood sample (20ml)
  Interventions: Procedure: Personalized Circulating DNA follow-up

INTERVENTIONS:
Procedure: Personalized Circulating DNA follow-up — FFPE tissue sample will be collected before and after surgery blood samples will be collected before and after surgery and every 3 to 4 months

SUMMARY:
PERCIMEL is an open multicentric study. The purpose of this study is to assess the interest of molecular analysis on circulating tumor DNA in the follow-up of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient;
* ECOG performance status 0-2;
* Patient with melanoma stage IIB or IIC, or any stage III, or stage IV that has been resected or is resectable;
* Treatment-naïve patient (except for initial excisional biopsy performed for diagnostic purposes);
* Patient scheduled to receive adjuvant therapy within 12 weeks following surgery, consisting of anti-BRAF and anti-MEK kinase inhibitors or anti-PD-1 monoclonal antibody immunotherapy, in accordance with marketing authorization;
* Patient with stage IIIB, IIIC, IIID, or IV melanoma with macroscopic lesions (clinically or radiologically detectable) eligible for neoadjuvant therapy, surgery, and adjuvant therapy (according to current recommendations: ESMO and NCCN guidelines, and treatment regimens from the SWOG S1801 and NADINA studies);
* Biological parameters compatible with the planned treatment;
* Patient informed and having provided written informed consent.

Exclusion Criteria:

* Patient with mucosal melanoma or choroidal (uveal) melanoma;
* Patient with another synchronous malignancy or who has been treated for another malignancy within the 3 years preceding informed consent (except carcinoma in situ of the cervix or resected cutaneous carcinoma);
* Contraindication to a 30 mL blood sample;
* Contraindication to surgery;
* Contraindication to the proposed medical treatment (anti-BRAF and anti-MEK targeted therapies or immunotherapy);
* Patient participating in another clinical trial involving an investigational medicinal product;
* Pregnant or breastfeeding woman;
* Patient deprived of liberty (including those under legal guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Studying the tumor molecular abnormalities resulting from circulating tumor DNA (ctDNA) to predict the resistance to treatment | 24 months
  Quantity of ctDNA / Resistance to treatment defined as a change in treatment decided during staff meeting

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU Jean Minjoz, Besançon
  - CGFL, Dijon
  - Chu Dijon, Dijon
  - Chru Lille, Lille
  - Ghr Mulhouse Sud Alsace, Mulhouse
  - Institut Godinot, Reims
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Chru Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No